CLINICAL TRIAL: NCT02821039
Title: Turkish Thoracic Society Usual Interstitial Pneumonia Registry Study
Acronym: TURK-UIP
Status: Terminated | Type: Observational
Why Stopped: We decided to complete our research in the 4th year, and publish the data. The data are under evaluation.
Sponsor: Turkish Thoracic Society (Other)
Responsible Party: Sponsor
Other Study IDs: TTS-01
Record Dates: First submitted 2016-06-29; First posted 2016-07-01 (Estimated); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Idiopathic Pulmonary Fibrosis; Usual Interstitial Pneumonia
Keywords: Idiopathic Pulmonary Fibrosis, Usual Interstitial Pneumonia
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The Turkish Thoracic Society Usual Interstitial Pneumonia Registry (TURK-UIP) is a collaborative project to coordinate a team of investigators from various regions of Turkey. The purpose of the Registry is to collect epidemiological data on patients with idiopathic pulmonary fibrosis and other causes of UIP, and to obtain information about the natural course of the disease and the treatment response.

DETAILED DESCRIPTION:
The TURK-UIP Registry is a web based application that will store information about patients. A HRCT pattern consistent with UIP will be confirmed by 3 radiologists. At the 3-month visits, the pulmonary function tests and the 6-minute walk test will be recorded. Patients will be prospectively followed for a 5-year period.

ELIGIBILITY:
Inclusion Criteria:

1. Understand and sign the informed consent document.
2. The presence of a definite or possible UIP pattern on high resolution computed tomography (HRCT) or a histologic UIP pattern (definite, probable and possible) on surgical lung biopsy (as defined by ATS/ERS/JRS/ALAT criteria).

Exclusion Criteria:

1. HRCT findings inconsistent with UIP pattern (peribronchovascular predominance, extensive ground glass abnormality,profuse micronodules, discrete cysts , consolidation in bronchopulmonary segment(s)/lobe(s), diffuse mosaic attenuation/air-trapping),
2. Histopathological findings inconsistent with UIP pattern (as defined by ATS/ERS/JRS/ALAT criteria).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects diagnosed with IPF and other causes of UIP.
Sampling Method: Non-Probability Sample
Enrollment: 1678 (Actual)
Dates: Start 2016-06; Primary Completion 2019-07-08 (Actual); Study Completion 2019-07-08 (Actual)

PRIMARY OUTCOMES:
Number of subjects enrolled with IPF and other causes of UIP | 5 years
  Natural history of course of disease in patients with IPF and other causes of UIP.

CONTACTS AND LOCATIONS:
Overall Officials: Benan Müsellim, MD, Principal Investigator — Istanbul University,Cerrahpasa Medical Faculty, Istanbul, Turkey.
Locations (45):
- Turkey (Türkiye) (45):
  - Cukurova University Medical Faculty, Adana
  - Sakarya University Faculty of Medicine, Adapazarı
  - Gazi University Medical Faculty, Ankara
  - Ankara University Faculty of Medicine, Ankara
  - Ankara University Medical Faculty, Ankara
  - Ataturk Chest Diseases and Chest Surgery Education and Research Hospital, Ankara
  - Atatürk Chest Disease and Chest Surgery Research and Training Hospital, Ankara
  - Dışkapı Yıldırım Beyazıt Training and Research Hospital, Ankara
  - Akdeniz University Medical Faculty, Antalya
  - Adnan Menderes University Faculty of Medicine, Aydin
  - Uludag University Medical Faculty, Bursa
  - Pamukkale University Medical Faculty, Denizli
  - Dicle University Medical Faculty, Diyarbakır
  - Memorial Diyarbakir Hospital, Diyarbakır
  - Duzce University Medical Faculty, Düzce
  - Trakya University Faculty of Medicine, Edirne
  - Atatürk University Faculty of Medicine, Erzurum
  - Atatürk University Medical Faculty, Erzurum
  - Dr.Lutfi Kirdar Kartal Education and Research Hospital, Istanbul
  - Istanbul University Cerrahpasa Medical Faculty, Istanbul
  - Istanbul University Istanbul Medical Faculty, Istanbul
  - Istanbul University, Istanbul Medical Faculty, Istanbul
  - Koç University Medical Faculty, Istanbul
  - Sisli Florence Nightingale Hospital, Istanbul
  - Sureyyapasa Chest Diseases and Thoracic Surgery Education and Research Hospital, Istanbul
  - Sureyyapasa Chest Diseases and Thoracic Surgery Training and Research Hospital, Istanbul
  - Süreyyapasa Pulmonary Diseases and Thoracic Surgery Education and Research Hospital, Istanbul
  - Yedikule Chest Disease Education and Research Hospital, Istanbul
  - Yedikule Chest Diseases and Chest Surgery Education and Research Hospital, Istanbul
  - Yedikule Chest Diseases and Thoracic Surgery Education and Research Hospital, Istanbul
  - Yedikule Chest Diseases Education and Research Hospital, Istanbul
  - Yedikule Hospital for Chest Disease and Chest Surgery, Istanbul
  - Yedikule Hospital for Chest Disease and Thoracic Surgery, Istanbul
  - Yedikule Pulmonary Diseases Education and Research Hospital, Istanbul
  - Dokuz Eylul University Medical Faculty, Izmir
  - Dr. Suat Seren Chest Diseases and Thoracic Surgery Training and Research Hospital, Izmir
  - Dr. Suat Seren Pulmonary Diseases and Thoracic Surgery Training and Research Hospital, Izmir
  - Ege University Faculty of Medicine, Izmir
  - Ege University Medical Faculty, Izmir
  - Kocaeli University Faculty of Medicine, Kocaeli
  - Kocaeli University Medical Faculty, Kocaeli
  - Necmettin Erbakan University Meram Medical Faculty, Konya
  - Kirikkale University Medical Faculty, Kırıkkale
  - Ondokuz Mayis University Medical Faculty, Samsun
  - Karadeniz Technical University Medical Faculty, Trabzon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Raghu G, Collard HR, Egan JJ, Martinez FJ, Behr J, Brown KK, Colby TV, Cordier JF, Flaherty KR, Lasky JA, Lynch DA, Ryu JH, Swigris JJ, Wells AU, Ancochea J, Bouros D, Carvalho C, Costabel U, Ebina M, Hansell DM, Johkoh T, Kim DS, King TE Jr, Kondoh Y, Myers J, Muller NL, Nicholson AG, Richeldi L, Selman M, Dudden RF, Griss BS, Protzko SL, Schunemann HJ; ATS/ERS/JRS/ALAT Committee on Idiopathic Pulmonary Fibrosis. An official ATS/ERS/JRS/ALAT statement: idiopathic pulmonary fibrosis: evidence-based guidelines for diagnosis and management. Am J Respir Crit Care Med. 2011 Mar 15;183(6):788-824. doi: 10.1164/rccm.2009-040GL. PMID 21471066
- [Background] American Thoracic Society; European Respiratory Society. American Thoracic Society/European Respiratory Society International Multidisciplinary Consensus Classification of the Idiopathic Interstitial Pneumonias. This joint statement of the American Thoracic Society (ATS), and the European Respiratory Society (ERS) was adopted by the ATS board of directors, June 2001 and by the ERS Executive Committee, June 2001. Am J Respir Crit Care Med. 2002 Jan 15;165(2):277-304. doi: 10.1164/ajrccm.165.2.ats01. No abstract available. PMID 11790668
- [Background] Ryerson CJ, Corte TJ, Collard HR, Richeldi L. A global registry for idiopathic pulmonary fibrosis: the time is now. Eur Respir J. 2014 Aug;44(2):273-6. doi: 10.1183/09031936.00051914. No abstract available. PMID 25082902